CLINICAL TRIAL: NCT01156194
Title: Effect of a Homeopathic Remedy on the Third Stage of Delivery: a Prospective, Randomized, Double-Blind Study.
Brief Title: Homeopathic Remedy for the Third Stage of Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ArBel.2010
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Third Stage of Labor
Keywords: third stage, labor, postpartum hemorrhage, homeopathy, arnica, bellis perennis
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Homeopathy 1 (Active Comparator): Arnica montana C6 and Bellis perennis C6
  Interventions: Drug: Homeopathy 1
- Homeopathy 2 (Active Comparator): Arnica montana C30 and Bellis perennis C30
  Interventions: Drug: Homeopathy 2
- Placebo (Placebo Comparator): globules identical to true comparators
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Homeopathy 1 — Arnica montana C6 and Bellis perennis C6
  Arms: Homeopathy 1
Drug: Homeopathy 2 — Arnica montana C30 and Bellis perennis C30
  Arms: Homeopathy 2
Drug: Placebo — globule identical to true homeopathy comparators
  Arms: Placebo

SUMMARY:
The homeopathic remedy consisting of Arnica and Bellis perennis have been shown in a previous pilot study (n=33) to reduce blood loss during the third stage of delivery, when compared with placebo treatment. The purpose of this study is to repeat the previous methodology, this time on a larger population.

210 parturients will be randomized to one of three groups: Arnica montana C6 and Bellis perennis C6 (n=70), Arnica montana C30 and Bellis perennis C30 (n=70), or double placebo (n=70).

ELIGIBILITY:
Inclusion Criteria:

* healthy women in 3rd stage of labor
* age 20-35
* second to fifth gestation
* spontaneous PV delivery
* term delivery (37-42nd weeks)

Exclusion Criteria:

* scarred uterus
* multifetal pregnancy
* history of bleeding problems
* caesarian section delivery
* chorioamnionitis
* pregnancy-induced hypertension
* gestational diabetes mellitus
* polyhydramnios, premature rupture of membrane
* suspected macrosomy/SGA

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin levels at 2d postpartum | 48h

SECONDARY OUTCOMES:
incidence of endometritis | 7d
time to extrusion of placenta following birth | 24h
duration of lochiae secretion | 7days
duration of third stage of labor | 24h
assessment of quality-of-life parameters | 7 days
assess toxic effects of the homeopathic remedies | 7 days
serum cortisol levels | within 12h postpartum
state of perineum postpartum | 48h

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Ward, Shaare Zedek Medical Center, Jerusalem, Israel